CLINICAL TRIAL: NCT02287857
Title: Efficacy and Safety of Domestic Tenofovir Tablets in Chinese Patients With Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTTQ-TDF-V4.0
Record Dates: First submitted 2014-10-30; First posted 2014-11-11 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Domestic Tenofovir Disoproxil Fumarate Tablets (Experimental)
  Interventions: Drug: Domestic Tenofovir Disoproxil Fumarate Tablets
- Tenofovir Disoproxil Fumarate Tablets of Gilead (Active Comparator)
  Interventions: Drug: Tenofovir Disoproxil Fumarate Tablets of Gilead

INTERVENTIONS:
Drug: Domestic Tenofovir Disoproxil Fumarate Tablets — 1 Domestic Tenofovir Disoproxil Fumarate Tablets and 1 blank Tenofovir Disoproxil Fumarate Tablets of Gilead
  Arms: Domestic Tenofovir Disoproxil Fumarate Tablets
Drug: Tenofovir Disoproxil Fumarate Tablets of Gilead — 1 blank Domestic Tenofovir Disoproxil Fumarate Tablets and 1Tenofovir Disoproxil Fumarate Tablets of Gilead
  Arms: Tenofovir Disoproxil Fumarate Tablets of Gilead

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Domestic Tenofovir Disoproxil Fumarate Tablets in Chinese patients with hepatitis B ,compared with Tenofovir Disoproxil Fumarate Tablets of Gilead.

ELIGIBILITY:
Inclusion Criteria:

* The initial treatment of subjects diagnosed of HBeAg positive or negative chronic hepatitis B
* Aged 18 to 65 years old，male or female
* Patients with previously HBsAg-positive lasted for 6months at least：HBeAg-positive subjects, HBV-DNA> 105copies/ml； HBeAg-negative subjects, HBV-DNA> 104copies/ml.
* 2 times the upper normal limit (2 × ULN) ≤ alanine aminotransferase (ALT) ≤ 10 × ULN.
* Total serum bilirubin (TBIL) ≤ 2.5 × ULN.
* Prothrombin activity (PTA) ≥ 60% or prothrombin time prolonged than normal ≤ 3 seconds).
* WBC ≥ 3.5 × 109 / L, PLT ≥ 80 × 109 / L, serum albumin (ALB)≥ 35 g / L.
* Creatinine (Cr) ≤ 1× ULN，serum phosphate was normal.
* Patients signed an informed consent form and compliance was good.

Exclusion Criteria:

* Patients were infected with other viruses as HAV, HCV, HEV, HIV etc.
* Patients with cirrhosis or liver cancer.
* Pregnant woman, lactating women .
* Patients with severe heart, kidney, endocrine hematopoietic system and neuropsychiatric diseases.
* Patients with metabolic or autoimmune diseases such as systemic lupus erythematosus.
* Patients allergic for study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Compared with baseline, decline of serum HBV-DNA in the value | 48 week

CONTACTS AND LOCATIONS:
Overall Officials: Yan yan Yu, doctor, Principal Investigator — Peking University First Hospital; Hao Wang, doctor, Principal Investigator — Peking University People's Hospital; Jun Chen, doctor, Principal Investigator — Beijing Ditan Hospital; Xin yue Chen, doctor, Principal Investigator — Beijing You An Hospital, Capital Medical University; Wen hong Zhang, doctor, Principal Investigator — Huashan Hospital; Qing Xie, doctor, Principal Investigator — Ruijin Hospital; Shan ming Wu, doctor, Principal Investigator — Shanghai Public Health Clinical Center; Hong Tang, doctor, Principal Investigator — West China Hospital; Qing Mao, doctor, Principal Investigator — First Affiliated Hospital, Third Military Medical University; Zhi liang Gao, doctor, Principal Investigator — Third Affiliated Hospital of Sun Yat-sen; Ji fang Shen, doctor, Principal Investigator — Zhejiang University; Jun Li, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Wei Zhao, doctor, Principal Investigator — The Second Hospital of Nanjing Medical University; Jia Shang, doctor, Principal Investigator — Henan Provincial People's Hospital; Zu jiang Yu, doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (15):
- China (15):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing You An Hospital, Capital Medical University, Beijing, Beijing Municipality
  - First Affiliated Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Third Affiliated Hospital of Sun Yat-sen, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdou, Sichuan
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Chen XF, Fan YN, Si CW, Yu YY, Shang J, Yu ZJ, Mao Q, Xie Q, Zhao W, Li J, Gao ZL, Wu SM, Tang H, Cheng J, Chen XY, Zhang WH, Wang H, Xu ZN, Wang L, Dai J, Xu JH. Tenofovir disoproxil fumarate in Chinese chronic hepatitis B patients: Results of a multicenter, double-blind, double-dummy, clinical trial at 96 weeks. World J Clin Cases. 2021 Jun 26;9(18):4690-4699. doi: 10.12998/wjcc.v9.i18.4690. PMID 34222435
- [Derived] Liang RY, Xu JH, Si CW, Wang S, Shang J, Yu ZJ, Mao Q, Xie Q, Zhao W, Li J, Gao ZL, Wu SM, Tang H, Cheng J, Chen XY, Zhang WH, Wang H, Xu ZN, Wang L, Dai J, Yu YY. A randomized, double-blind, double-dummy, controlled, multicenter study of Qingzhong (tenofovir disoproxil fumarate) versus Viread for the treatment of chronic hepatitis B: First-stage results at week 48. Medicine (Baltimore). 2019 Aug;98(33):e16778. doi: 10.1097/MD.0000000000016778. PMID 31415381